CLINICAL TRIAL: NCT06435221
Title: A Multicenter, Open-Label Study Assessing Long-Term Exposure With Cytisinicline 3 mg TID
Brief Title: Safety Study of Cytisinicline in Adult Combustible and/or E-cigarette Smokers
Acronym: ORCA-OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-13
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Vaping Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cytisinicline 3 mg TID (Experimental): Cytisinicline 3 mg TID for 52 weeks.
  Interventions: Drug: Cytisinicline

INTERVENTIONS:
Drug: Cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: Cytisine

SUMMARY:
Safety assessment of long-term 3 mg cytisinicline three times daily (TID) exposure for 52 weeks is the main purpose of this study, conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Prior participation in the ORCA-2, ORCA-3 or ORCA-V1 clinical studies.
2. Former ORCA-2/ORCA-3 and ORCA-V1 subjects who are current daily cigarette smokers and/or daily nicotine-containing electronic cigarette users. Amount of daily combustible and/or nicotine containing electronic cigarette use at baseline is determined by subject self-report.
3. At Screening, subjects must have expired carbon monoxide (CO) ≥10 ppm if self-reporting as smokers or ≥30 ng/mL cotinine using a point-of-care cotinine oral fluid screening device if self-reporting as users of nicotine containing electronic cigarettes.
4. Willing to initiate cytisinicline treatment on the day after enrollment and set a quit date within 14 days of starting treatment.
5. Willing to actively participate in the study's cessation behavioral support provided throughout the study.
6. Able to fully understand study requirements, willing to participate, and comply with dosing schedule.
7. Sign the Informed Consent Form.

Exclusion Criteria:

1. Known hypersensitivity to cytisinicline or any of the excipients.
2. Clinically significant abnormal screening serum chemistry or hematology values.
3. Clinically significant abnormal screening 12-lead ECG determined after minimum of 5 minutes in supine position (ie, requiring treatment or further assessment).
4. Recent history (within 3 months prior to screening) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident or hospitalization for congestive heart failure.
5. Current uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg).
6. Currently psychotic or having had a psychotic event within 3 months prior to screening; currently having suicidal ideation or risk for suicide (corresponding to question 4 or 5 on the screening C-SSRS OR "Yes" to any suicidal behavior question on the screening C-SSRS with clear suicidal intent or previous attempt); or current symptoms of moderate to severe depression (depression score ≥11 on the HADS) at screening. If any subject becomes psychotic during the study, they must be removed from cytisinicline treatment and/or additional study visits.
7. Severe renal impairment defined as a creatinine clearance (CrCl) <60 mL/min on screening lab (estimated with the Cockroft-Gault equation).
8. Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 x the upper limit of normal (ULN) on screening lab.
9. Women who are pregnant or breast-feeding.
10. Female subjects of childbearing potential who do not agree to use acceptable methods of birth control during the study. Acceptable methods of birth control include:

    * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
    * Barrier methods:

      * diaphragm
      * cervical cap
      * contraceptive sponge
    * Hormonal methods:

      * Oral contraceptives
      * Vaginal ring such as NuvaRing
      * Skin patch such as Xulane
      * Injection such as Depro-Provera
      * Implantable rod such as Nexplanon
11. Participation in a clinical study with an investigational drug in the 4 weeks prior to enrollment.
12. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Treatment Emergent Serious Adverse Events (SAEs) | up to Week 52

SECONDARY OUTCOMES:
Incidence Rate of Related Treatment Emergent SAEs | up to Week 52
Incidence Rate of Treatment Emergent Adverse Events (TEAEs) | up to Week 52
Incidence Rate of Related TEAEs | up to Week 52
Number of Participants With Clinically Significant Abnormal Hematology and Chemistry Parameters | up to Week 52
Percentage of Participants With Clinically Significant Abnormal Hematology and Chemistry Parameters | up to Week 52
Number of Participants With Potentially Clinically Significant Abnormal Vital Signs | up to Week 52
Percentage of Participants With Potentially Clinically Significant Abnormal Vital Signs | up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ball, Study Director — Achieve Life Sciences, Inc.
Locations (29):
- United States (29):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Little Rock Allergy & Asthma Clinical Research Center, Little Rock, Arkansas
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Accel Research Sites Network - DeLand Clinical Research Unit, DeLand, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Alliance for Multispecialty Research, LLC, Oak Brook, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Massachusetts General Hospital - Clinical Genetic Facility, Boston, Massachusetts
  - Insight Research Institute, Flint, Michigan
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Global Medical Institutes LLC; Princeton Medical Institute, Princeton, New Jersey
  - Rochester Clinical Research, LLC, Rochester, New York
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No